CLINICAL TRIAL: NCT01089803
Title: Observational Study of Swallowing Function After Treatment of Advanced Laryngeal Cancer
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other); American Head and Neck Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2008NTLS104; 0809M45481 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Squamous Cell Carcinoma; Laryngeal Cancer
Keywords: laryngectomy; larynx; hypopharynx
MeSH Terms: conditions — Carcinoma, Squamous Cell; Laryngeal Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients Treated with Laryngectomy: Patients initially treated with laryngectomy and followed for 12 months after receiving this treatment.
- Patients Treated with Chemoradiation: Patients treated initially with chemoradiation and followed for 12 months after receiving treatment.

SUMMARY:
The purpose of this prospective, multi-institutional, observational cohort study is to determine if an initial surgical approach leads to better function and quality of life than primary chemoradiation in a subset of patients with advanced hypopharyngeal and laryngeal cancers.

DETAILED DESCRIPTION:
At the time of registration patients will be categorized into 2 groups based on the initial treatment plan as either chemoradiation-based or surgically-based (laryngectomy). Treatment will be assigned by the patient's physician, it will not be assigned by the study.

Patients will be asked to complete a series of 4 questionnaires addressing swallowing function, generic health status, head and neck cancer-specific quality of life, and self-reported speech function at 3 time points (baseline, 6 months and 12 months after the end of treatment). The treating physician will provide basic clinical information at these same time points. In centers where swallowing and voice assessments are done as part of standard of care, data from these studies will also be provided.

Study entry is open to all adults regardless of gender or ethnic background. Specific information regarding the definitive treatment (surgery or chemoradiation) will be provided to the patient by the treating physician as part of the routine standard of care. Any treatment related side effects, as well as the duration of therapy and follow-up will be managed by the treating physician. Participation in this study will have no effect on the initial treatment decisions or the course of care.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to complete self-administered follow-up questionnaires over the course of one year as determined by a member of the research team
* Voluntary written informed consent with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Must be at least 18 years of age

Exclusion Criteria:

* Require a resection that would involve more than the standard laryngectomy (total pharyngectomy, esophagectomy)
* Undergo partial laryngectomy, when open or endoscopic
* Have previously altered anatomy of the upper aerodigestive tract
* Have pre-existing dysphagia unrelated to the tumor, or neurologic disorders that could affect swallowing (Parkinson's, cerebrovascular accidents)
* Have prior malignant disease of the upper aerodigestive tract
* Have prior radiation therapy to the head and neck region
* Metastatic disease
* Unable to complete self-administered questionnaires written in simple English for cognitive, psychiatric, or other reasons that in the opinion of the enrolling investigator is likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed squamous cell carcinoma of the larynx (cartilage invading-T3 and all T4) or hypopharynx (T2 and T3) for which curative treatment is planned. The tumor must be resectable with total laryngectomy alone as determined by the treating surgeon - this requirement is regardless of whether the surgery of chemoradiation is planned for the patient.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2009-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Swallowing Function Scores | 12 months after Treatment
  The primary outcome will be self-reported swallowing function (M.D. Anderson Dysphagia Inventory questionnaire - MDADI) 12 months after treatment. Analysis will compare MDADI scores of patients treated initially with laryngectomy vs. those of patients treated initially with chemoradiation.

SECONDARY OUTCOMES:
General Quality of Life | PreTreatment, 6 Months and 12 Months After Treatment
  The SF-12 Quality of Life questionnaire will be used to assess general health status. The SF-12 contains one or two items that measure each of eight domains of health: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It yields scale scores for each of these eight health domains, and two summary measures of physical and mental health: the Physical Component Summary (PCS) and Mental Component Summary (MCS).
Speech Assessment | PreTreatment, 6 Months and 12 Months After Treatment
  Speech analysis will focus primarily on speech intelligibilty and acceptability to both clinicians and naive listeners, and less on voice quality per se using the Voice Handicap Index. The Voice Handicap Index (VHI) measures the influence of voice problems on a patient's quality of life.
Head and Neck Quality of Life | PreTreatment, 6 Months and 12 Month After Treatment
  The University of Washington Quality of Life Assessment Questionnaire will be administered. This questionnaire is specifically designed to capture head and neck cancer-specific function.

CONTACTS AND LOCATIONS:
Overall Officials: Bevan Yueh, MD, MPH, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States